CLINICAL TRIAL: NCT05020938
Title: Long Term Follow-Up of KNEE PAIN Patients Accompanying Meniscus Tear Treated With Integrated Complementary and Alternative
Brief Title: Long Term Follow-Up of KNEE PAIN Patients Accompanying Meniscus Tear
Status: Completed | Type: Observational
Sponsor: Jaseng Medical Foundation (Other)
Responsible Party: Principal Investigator, In-Hyuk Ha, KMD, Director, Jaseng Medical Foundation
Other Study IDs: JS-CT-2021-12
Record Dates: First submitted 2021-08-23; First posted 2021-08-25 (Actual); Last update posted 2022-01-14 (Actual); Status verified 2022-01

CONDITIONS: Meniscus Tear

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: phone survey — A questionnaire about the current symptoms and satisfaction for received treatment will be conducted over the phone for patients.

SUMMARY:
The purpose of this study is to reveal the effectiveness and satisfaction of integrative Korean medicine for Meniscus Tear by observation patients treated with integrative Korean medicine.

This study is a prospective observational study. The subjects for study are patients diagnosed with Meniscus Tear and who have been admitted to Gangnam Jaseng Hospital of Korean medicine, Bucheon Jaseng Hospital of Korean medicine, Daejeon Jaseng Hospital of Korean medicine and Haeundae Jaseng Hospital of Korean medicine for 2015.06-2020.06.

DETAILED DESCRIPTION:
Medical records of selected patients will be analyzed, and telephone surveys will be conducted for each patient. The survey questions are Numeric rating scale (NRS), Western Ontario and McMasters Universities(WOMAC) Osteoarthritis Index, quality of life, and Patient Global Impression of Change (PGIC), etc.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who have been diagnosed with "Meniscus Tear" in the EMR imaging (X-ray or MRI or CT) of hospitalization
2. Patients who have been hospitalized by Knee Pain
3. A person who voluntarily orally agrees to participate in a clinical trial

Exclusion Criteria:

1. If the hospitalization period is less than 3 days,
2. If there are other chronic diseases that may interfere with the treatment effect or interpretation of the results: cardiovascular disease, kidney disease, diabetic neuropathy, dementia, epilepsy, etc.
3. If the cause of pain is caused by a soft tissue disease other than Knee joint: tumor, fibromyalgia, rheumatoid arthritis, gout, etc.
4. Patients within 3 months of surgery on the hip joint
5. If there is a fracture of the joint in the image finding
6. If researchers judge that it is inappropriate to participate in the study;
7. If you do not agree to participate in the study;
8. Minors

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The target is those who showed Meniscus Tear in video findings among patients admitted to Gangnam Mainwon, Daejeon, and Bucheon Haeundae, four branches of Hospitals with Knee pain from June 2015 to June 30, 2020.
Sampling Method: Non-Probability Sample
Enrollment: 86 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-11-15 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
Numeric Rating Scale (NRS) | Finish survey by August 2021
  NRS uses an 11-point scale to evaluate current knee pain where no pain is indicated by '0', and the worst pain imaginable by '10'. NRS was assessed at admission, 2 weeks after admission, discharge, and long term follow up.

SECONDARY OUTCOMES:
Western Ontario and McMasters Universities(WOMAC) Osteoarthritis Index | Finish survey by August 2021
  Knee Pain intensity scale
EuroQol 5 Dimension (EQ 5D 5L) | Finish survey by August 2021
  5 Level Quality of life
Patient Global Impression of Change (PGIC) | Finish survey by August 2021
  PGIC is an indicator that evaluates the improvement of patients in 5 steps, and the subject responds with improvement of functional limitation after treatment with 5 likert. (1=completely improved, 2=distinctly improved, 3=improved, 4=no significant difference, 5=worsened)

CONTACTS AND LOCATIONS:
Overall Officials: In-Hyuk Ha, Ph.D, Study Director — Jaseng Medical Foundation
Locations (1):
- Jaseng Hospital of Korean Medicine, Seoul, Gangnam-Gu, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lee JH, Song JY, Park KS, Lee J, Ha IH, Lee YJ. Long-term follow-up of inpatients with meniscus tears who received integrative Korean medicine treatment: A retrospective analysis and follow-up survey. Medicine (Baltimore). 2024 Feb 9;103(6):e36917. doi: 10.1097/MD.0000000000036917. PMID 38335386